CLINICAL TRIAL: NCT01394120
Title: Phase II Study of Chemotherapy Selection Based on Therapeutic Targets for the Treatment of Advanced Pancreatic Cancer
Brief Title: Chemotherapy Selection Based on Therapeutic Targets for Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sofia Perea, Director Clinical Trials Unit. (Other)
Responsible Party: Sponsor-Investigator, Sofia Perea, Director Clinical Trials Unit., Director Clinical Trial Unit, Grupo Hospital de Madrid
Organization: Grupo Hospital de Madrid (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARGTHPANC 001; 2011-001017-13 (EudraCT Number)
Record Dates: First submitted 2011-07-05; First posted 2011-07-14 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Pancreas cancer; Targeted Therapy
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tarteted Therapy (Experimental)
  Interventions: Drug: Targeted Therapy Tailored Treatment
- Standard Chemotherapy (Active Comparator)
  Interventions: Drug: Standard Chemotherapy

INTERVENTIONS:
Drug: Targeted Therapy Tailored Treatment — Targeted therapy tailored treatment, based on molecular determination in pancreas cancer specimen
  * Tim Synthase (TS) (neg), ERCC-1 (neg), Topoisomerase I (Topo I) (pos) : FOLFIRINOX
  * TS (neg), ERCC-1 (neg), Topo I (neg): FOLFOX
  * TS (neg), ERCC-1 (pos), Topo I (pos): FOLFIRI
  * TS (neg), ERCC-1 (pos), Topo I (neg): Capecitabine/Gemcitabine
  * TS (pos), EGFR Not Amplificate, K-Ras Mutation (pos) : Gemcitabine single agent
  * TS (pos), EGFR Ampl or K-Ras mut (neg): Gemcitabine plus Erlotinib
  Other Names: Individualized treatment selection based on predictors of response biomarkers
  Arms: Tarteted Therapy
Drug: Standard Chemotherapy — Patients treated based on investigator´s criteria: : FOLFIRINOX, FOLFOX, FOLFIRI, Capecitabine-Gemcitabine, Erlotinib-Gemcitabine or Gemcitabine single agent
  Other Names: Treatment at the investigator's discretion
  Arms: Standard Chemotherapy

SUMMARY:
In recent years, treatment of advanced pancreatic cancer is changing. Currently, there are several active schedules of chemotherapy that can be used, such as gemcitabine as monotherapy or in combination with capecitabine or erlotinib, and FOLFIRINOX. Moreover, the development of biomarker (therapeutic targets) that can predicte response to treatment is a new important tool to be used in clinical practice to select the best scheme for each patient. Preliminary studies showed that therapeutic target determination, using tumor tissue collected from patients, could determine the presence of groups of "chemotherapy responders". Such is the case of EGFR amplification and/or K-Ras gene status and correlation with response to erlotinib. Moreover, Thymidilate Synthase, Thimidine Phosphorylase, ERCC-1 and Topoisomerase I expression by immunohistochemistry in GI tumor samples has been related to resistance or response to 5FU-capecitabine, oxaliplatin and irinotecan respectively. Based on this data the investigators designed a phase II clinical trial to evaluate the efficacy of selected treatment for pancreatic cancer patients based on the determination of therapeutic targets. The therapeutic target-driven treatment efficacy will be compared to the prospective treatment of a control group of patients treated at the discretion of the physician-researcher

DETAILED DESCRIPTION:
Study Phase: Phase 2 Trial

Study Objetives:

* Primary end-point. Proportion of patients alive after 12 months in patients with advanced pancreatic carcinoma individually selected and grouped according to the expression in tumor tissue for therapeutic targets.
* Secondary end-points. 1. Assessing the feasibility of the method of patient-treatment-selection based on tumor tissue expression of therapeutic targets. 2. Overal survival comparison between Gemcitabine single agent treatment and the rest of chemotherapy schedules. 3. Determination of progression-free survival for each treatment group. 4. Determination of toxicity in all the patients.

Study population and Number of subject: A total of 60 pancreatic cancer patients with advanced pancreas cancer with no previous systemic treatment are expected to be enrolled.

Study design and schedule. Patients will be randomized (1:1) to a control arm or an experimental treatment arm guided by therapeutic targets. In the control arm, patients are treated with conventional chemotherapy regimens at the discretion of the investigator. In the experimental arm, patients are treated as determined in tumor tissue available for biomarker TS, TP, ERCC-1, Topo-1, K-Ras mutation and EGFR FISH, choosing FOLFIRINOX schemas, FOLFOX, FOLFIRI, Gemcitabine-Capecitabine Gemcitabine-Erlotinib, Gemcitabine single agent. All patients will be analyzed by intention to treat

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of pancreas adenocarcinoma
* Clinical stage IV
* Feasible patient for chemotherapy
* Availability of tumor tissue or possibility of a tumor biopsy to define therapeutic targets
* Informed written consent

Exclusion Criteria:

* Previous systemic treatment for advanced pancreas adenocarcinoma
* Contraindication to the administration of any of the drugs used in the study: capecitabine, 5Fluouracil, irinotecan, oxaliplatin, gemcitabine or erlotinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, Principal Investigator
Locations (1):
- Centro Integral Oncologico Clara Campal, Madrid, Spain